CLINICAL TRIAL: NCT05608772
Title: Conversion of Failed Sleeve Gastrectomy Due to Weight Regain to SADI-S, RYGB or OAGB
Brief Title: Conversion to SADI-S, RYGB or OAGB After Failed Sleeve
Acronym: RCTresleeve
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Mohamed Hany Ashour, ass professor, General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT-revision-3arms
Record Dates: First submitted 2022-10-25; First posted 2022-11-08 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Weight Loss; Bariatric Surgery Candidate; Comorbidities and Coexisting Conditions; Nutrient Deficiency
Keywords: RYGB; OAGB; SADI-S; Sleeve gastrectomy
MeSH Terms: conditions — Weight Loss | interventions — Reoperation

STUDY DESIGN:
Intervention Model Description: A single-blind randomization procedure, in which patients and outpatient clinic nurses will be blinded to the study period p
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RYGB procedure arm 1 (Active Comparator): After failed sleeve, the patients will get a revisional procedure. The RYGB
  Interventions: Procedure: revision surgery
- OAGB procedure arm 2 (Active Comparator): After failed sleeve, the patients will get a revisional procedure. The OAGB
  Interventions: Procedure: revision surgery
- SADI-S procedure arm 3 (Active Comparator): After failed sleeve, the patients will get a revisional procedure. The SADI-S
  Interventions: Procedure: revision surgery

INTERVENTIONS:
Procedure: revision surgery — revision procedure after failed sleeve gastrectomy

SUMMARY:
Assess what revisional surgery is superior and provides the best weight loss after primary LSG. What is the occurrence of complications and the nutritional laboratory status? And if the resolution and /or improvement of associated medical problems after the weight loss will occur.

DETAILED DESCRIPTION:
Laparoscopic sleeve gastrectomy (LSG) gained popularity and has become one of the most performed weight loss procedures worldwide. In the long-term follow-up, the literature states that the incidence of gastroesophageal reflux disease (GERD) accounts for 16%, and weight regains accounting for 70% after LSG. These are the two most common complications which can necessitate further surgical intervention.

The hypotheses are that laparoscopic conversion from LSG to Single anastomosis duodeno-ileal bypass (SADI-S), Roux-en-Y gastric bypass (RYGB), or one anastomosis gastric bypass (OAGB) will provide a new significant weight loss, improvement in obesity-related health problems and provide no nutritional deficiency in all cases.

Since the three types of procedures have other anatomical presentations, whereby these is not well tested next to each other in a blinded, controlled setting for the patient, this study is designed to discover if the procedures are superior to each other or not and what the best outcome is for the patient.

A sample size is calculated and with a medium effect size of 0.5 corresponds to a mean difference in %EBMIL between SADI-S, RYGB, and OAGB of at least 10%. Using a power of 0.8 with an alpha of 0.05 resulted in a sample size of 64 patients per group.

Considering a possible loss of patients to follow-up, an additional 20% increase in sample size was included per group, resulting in a minimum of 78 patients per group.

(Total of 3 groups together of 234 patients).

ELIGIBILITY:
Inclusion Criteria:

* Undergone primary laparoscopic sleeve gastrectomy in the past
* Weight regain

  * defined as any increase in weight above the nadir as reported by the patient
  * BMI at the time of revisional surgery was around 45 kg/m2
  * weight regain was defined as an increase in BMI after bariatric surgery to exceed 35
* With or without Gastroesophageal reflux disease (GERD) grade A and B o Patients with grade C or higher GERD, according to the Los Angeles (LA) classification [7] will be excluded from the study

Exclusion Criteria:

* Didn't follow preoperative consultation
* Cannot give of sign informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 234 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2028-03-15 (Estimated); Study Completion 2028-04-15 (Estimated)

PRIMARY OUTCOMES:
The number of participants who will have early complications related to surgery | 6 weeks
  the incidence of re-operation, bleeding or leakages
The percentage Excess body weight loss (%EWL) | 3,6,12,24 months
  the amount of weight loss after revision surgery
somscore of food tolerance | 2,6 weeks and 3,6,12,24 months
  validated food tolerance questions: Food tolerance (FT) was evaluated using a one-page questionnaire divided into 4 sections, 3 of which were used to calculate the score: overall patient satisfaction with eating (score: 1-5); tolerability to certain food types (score: 0-16); and frequency of vomiting/regurgitation (score: 0-6), with a total score between 1 and 27; higher scores indicate better food tolerance

SECONDARY OUTCOMES:
Nutritional levels of albuminemia | 3,6,12,24 months
  the albuminemia level will be tested after surgery (g/dl)
Nutritional levels of proteinemia | 3,6,12,24 months
  the proteinemia level will be tested after surgery (mg/dl)
Nutritional levels of anemia | 3,6,12,24 months
  the anemia level will be tested after surgery (Mcl)
Nutritional levels of calcemic | 3,6,12,24 months
  the calcemic level will be tested after surgery (mg/dl)
Incidence of Reflux | 3,6,12,24 months
  GERD assessment
The number of participants who will have late complications related to surgery | 3,6,12,24 months
  the incidence of re-operations will be collected
Short Form 36 Quality of life | 3,6,12,24 months
  Quality of life assessment will be tested 8 chapters with in total 36 questions and a somscore from 0-100 will be calculated (the higher the somscore the better the quality of life is).
VAS/NRS (incidence of pain) | 3,6,12,24 months
  pain scoring from 0-10 (0 is no pain 10 is most worst pain)
Metabolic biomarkers Glucagon-like peptide-1 (GLP1) | 3,6,12,24 months
  the GLP1 level will be tested after surgery (mg/ml)
Metabolic biomarkers Leptin | 3,6,12,24 months
  the Leptin level will be tested after surgery (mg/ml)
Metabolic biomarkers Peptide YY ( PYY) | 3,6,12,24 months
  the PYY level will be tested after surgery (pg/ml)
Metabolic biomarkers Ghrelin | 3,6,12,24 months
  the Ghrelin level will be tested after surgery (mg/ml)
Metabolic biomarkers Insulin | 3,6,12,24 months
  the Insulin level will be tested after surgery (million units/ml)

OTHER OUTCOMES:
The number of participants who will have late complications related to surgery | 60 months
  the incidence of re-operations or complications will be collected
The number of participants whereby revision surgery necessary after the RCT | 60 months
  the incidence of re-operations or other procedure will be collected
The percentage Excess body weight loss (%EWL) | 60 months
  the amount of weight loss after revision surgery
Incidence of Reflux | 60 months
  GERD classification
Nutritional levels of albuminemia | 60 months
  the albuminemia level will be tested after surgery (g/dl)
Nutritional levels of proteinemia | 60 months
  the proteinemia level will be tested after surgery (mg/dl)
Nutritional levels of anemia | 60 months
  the anemia level will be tested after surgery (Mcl)
Nutritional levels of calcemic | 60 months
  the calcemic level will be tested after surgery (mg/dl)
Somscore of food tolerance | 60 months
  validated food tolerance questions: Food tolerance (FT) was evaluated using a one-page questionnaire divided into 4 sections, 3 of which were used to calculate the score: overall patient satisfaction with eating (score: 1-5); tolerability to certain food types (score: 0-16); and frequency of vomiting/regurgitation (score: 0-6), with a total score between 1 and 27; higher scores indicate better food tolerance
Short Form 36 Quality of life | 60 months
  Quality of life assessment will be tested 8 chapters with in total 36 questions and a somscore from 0-100 will be calculated (the higher the somscore the better the quality of life is).
VAS/NRS (incidence of pain) | 60 months
  pain scoring from 0-10 (0 is no pain 10 is most worst pain)
Metabolic biomarkers Glucagon-like peptide-1 (GLP1) | 60 months
  the GLP1 level will be tested after surgery (mg/ml)
Metabolic biomarkers Leptin | 60 months
  the Leptin level will be tested after surgery (mg/ml)
Metabolic biomarkers Peptide YY ( PYY) | 60 months
  the PYY level will be tested after surgery (pg/ml)
Metabolic biomarkers Ghrelin | 60 months
  the Ghrelin level will be tested after surgery (mg/ml)
Metabolic biomarkers Insulin | 60 months
  the Insulin level will be tested after surgery (million units/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ashour, MD, Principal Investigator — University of Alexandria
Locations (1):
- Madina Women's Hospital, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
FAIR data of this study can be requested. All will be saved in the Castor Electronic data capture system.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After 2 and 5 years and after full analysis and publication the data will be available and stored for minimal 10 years.
Access Criteria: Email the Principal investigator. Whereby access to an annonymous database site will be created.

REFERENCES:
- [Background] Guan B, Chong TH, Peng J, Chen Y, Wang C, Yang J. Mid-long-term Revisional Surgery After Sleeve Gastrectomy: a Systematic Review and Meta-analysis. Obes Surg. 2019 Jun;29(6):1965-1975. doi: 10.1007/s11695-019-03842-3. PMID 30903425
- [Background] Lazzati A, Bechet S, Jouma S, Paolino L, Jung C. Revision surgery after sleeve gastrectomy: a nationwide study with 10 years of follow-up. Surg Obes Relat Dis. 2020 Oct;16(10):1497-1504. doi: 10.1016/j.soard.2020.05.021. Epub 2020 May 29. PMID 32636173
- [Background] Clapp B, Wynn M, Martyn C, Foster C, O'Dell M, Tyroch A. Long term (7 or more years) outcomes of the sleeve gastrectomy: a meta-analysis. Surg Obes Relat Dis. 2018 Jun;14(6):741-747. doi: 10.1016/j.soard.2018.02.027. Epub 2018 Mar 6. PMID 29625744
- [Background] Parmar CD, Gan J, Stier C, Dong Z, Chiappetta S, El-Kadre L, Bashah MM, Wang C, Sakran N. One Anastomosis/Mini Gastric Bypass (OAGB-MGB) as revisional bariatric surgery after failed primary adjustable gastric band (LAGB) and sleeve gastrectomy (SG): A systematic review of 1075 patients. Int J Surg. 2020 Sep;81:32-38. doi: 10.1016/j.ijsu.2020.07.007. Epub 2020 Jul 29. PMID 32738545
- [Background] Chiappetta S, Stier C, Scheffel O, Squillante S, Weiner RA. Mini/One Anastomosis Gastric Bypass Versus Roux-en-Y Gastric Bypass as a Second Step Procedure After Sleeve Gastrectomy-a Retrospective Cohort Study. Obes Surg. 2019 Mar;29(3):819-827. doi: 10.1007/s11695-018-03629-y. PMID 30542828
- [Background] Angrisani L, Santonicola A, Iovino P, Ramos A, Shikora S, Kow L. Bariatric Surgery Survey 2018: Similarities and Disparities Among the 5 IFSO Chapters. Obes Surg. 2021 May;31(5):1937-1948. doi: 10.1007/s11695-020-05207-7. Epub 2021 Jan 12. PMID 33432483
- [Background] Sami S, Ragunath K. The Los Angeles Classification of Gastroesophageal Reflux Disease. Video Journal and Encyclopedia of GI Endoscopy. 2013;1:103-4.